CLINICAL TRIAL: NCT06961864
Title: Visual Perception in Visual Snow Syndrome
Brief Title: Investigating Brain Function in People With and Without Visual Snow Syndrome Using Adaptation to Visual Stimuli
Acronym: VPVSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Mayo Clinic (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00014113; R01EY036005 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Visual Snow Syndrome; Migraine; Healthy
Keywords: Visual Snow Syndrome; Visual Snow; Migraine; Floaters; Palinopsia; Photophobia; Nyctalopia; Entoptic phenomena; Visual trailing; Adaptation; Magnetic resonance spectroscopy; MRS; Magnetic resonance imaging; MRI; University of Minnesota; Afterimages; Poor night vision; Light sensitivity; Persistent positive visual phenomena; Static
MeSH Terms: conditions — visual snow syndrome; Migraine Disorders; vitreous floaters; palinopsia; Photophobia; Night Blindness; Vitamin A Deficiency | interventions — Surveys and Questionnaires; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with Visual Snow Syndrome (Active Comparator)
  Interventions: Behavioral: Visual Adaptation; Behavioral: Assessments and Questionnaires; Device: Functional Magnetic Resonance Imaging (fMRI); Device: Magnetic Resonance Imaging (MRS)
- Non-snow Controls (Placebo Comparator)
  Interventions: Behavioral: Visual Adaptation; Behavioral: Assessments and Questionnaires; Device: Functional Magnetic Resonance Imaging (fMRI); Device: Magnetic Resonance Imaging (MRS)

INTERVENTIONS:
Behavioral: Visual Adaptation — Presentation of visual stimuli to quantify the appearance of visual snow or its effects in the visual system of the brain.
Behavioral: Assessments and Questionnaires — Administration of clinical assessments and questionnaires to gather information about visual and mental symptoms, cognitive, and sensory function.
Device: Functional Magnetic Resonance Imaging (fMRI) — 7 tesla fMRI data will be acquired during visual paradigms designed to measure neural responses with and without adaptation.
Device: Magnetic Resonance Imaging (MRS) — 7 tesla MRS data will be acquired to quantify the concentrations of different brain chemicals in brain regions including visual cortex.

SUMMARY:
The goal of this study is to learn more about the brain pathways and activity involved in creating Visual Snow Syndrome (VSS). The main questions it aims to answer are:

* Does VSS arise from spontaneous activity in brain pathways?
* Where in the brain does the activity contributing to VSS arise?
* How does brain activity contribute to VSS?

Participants will:

1. Undergo assessments and questionnaires to understand visual and mental symptoms, cognitive, and sensory function.
2. Make visual judgements based on images presented to them both inside and outside a magnetic resonance imaging (MRI) machine.
3. Undergo scanning of their brain while inside of an MRI machine.

ELIGIBILITY:
Inclusion Criteria for People with Visual Snow Syndrome:

* Between the ages of 18 and 60 years old
* Normal (20/25 or better in each eye) or corrected-to-normal vision (MR-compatible glasses will be provided as needed)
* Ability to comply with study instructions
* Individuals who have a current diagnosis of VSS from a neuro-ophthalmologist or meet diagnostic criteria of VSS (experience of dynamic dots across the visual field persisting longer than 3 months and at least 2 of the following additional visual symptoms: palinopsia, entoptic phenomena, trails behind moving objects, photophobia, or nyctalopia)
* Individuals living in Minnesota within 2 hours of the study site

Inclusion Criteria for Non-snow Controls:

* Between the ages of 18 and 60 years old
* Normal (20/25 or better in each eye) or corrected-to-normal vision (MR-compatible glasses will be provided as needed)
* Ability to comply with study instructions
* Individuals living in Minnesota within 2 hours of the study site

Exclusion Criteria for People with Visual Snow Syndrome:

* Not being fluent in English or another language for which interpretation/translation services are available
* A diagnosed or self-reported intellectual disability
* Current substance dependence (besides nicotine), or drug dependence with tolerance or withdrawal within past 12 months
* Hallucinogenic substance use within the past 12 months or hallucinogenic substance use within 12 months prior to onset of VSS symptoms
* Severe central nervous system disease
* Head injury with skull fracture or loss of consciousness for more than thirty minutes
* Presence of a physical problem that would render study measures difficult or impossible to administer or interpret (e.g., visual field loss)
* Age less than 18 years or greater than 60 years
* MRI exclusions (for MR visits only):

  * Metal in the body that cannot be approved by the CMRR safety committee
  * Pregnancy
  * Conditions that affect neuro-hemodynamic coupling
  * Claustrophobia
  * Inability to lie still for at least an hour
  * Weight in excess of 440 lbs
  * CT scan exclusion only: Research-related radiation exposure within the last 12 months
* Any vision anomaly aside from VS or refractive error (e.g., strabismus/ crossed eyes, lazy eyes, color blindness)
* Current psychotic episode

Exclusion Criteria for Non-snow Controls:

* Not being fluent in English or another language for which interpretation/translation services are available
* A diagnosed or self-reported intellectual disability
* Current substance dependence (besides nicotine), or drug dependence with tolerance or withdrawal within past 12 months
* Hallucinogenic substance use within the past 12 months
* Severe central nervous system disease
* Head injury with skull fracture or loss of consciousness for more than thirty minutes
* Presence of a physical problem that would render study measures difficult or impossible to administer or interpret (e.g., visual field loss)
* Age less than 18 years or greater than 60 years
* MRI exclusions (for MR visits only):

  * Metal in the body that cannot be approved by the CMRR safety committee
  * Pregnancy
  * Conditions that affect neuro-hemodynamic coupling
  * Claustrophobia
  * Inability to lie still for at least an hour
  * Weight in excess of 440 lbs
  * CT scan exclusion only: Research-related radiation exposure within the last 12 months
* Any vision anomaly or refractive error (e.g. strabismus/ crossed eyes, lazy eyes, color blind)
* A personal history of VSS symptoms or a diagnosis with VSS
* Current psychotic episode

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Psychophysical Adaptation Task Performance | 1.5-2 hours per session, with experiments divided across multiple (e.g., 3) sessions
  Visual tasks will consist of perceptual judgments following adaptation (e.g., subject will report when internal or external / simulated visual snow appears the same on the left or right side of the screen). Measures will be compared for visual target stimuli in different task conditions and experiments, with the goal of understanding the neural basis of visual snow.
Functional Magnetic Resonance Imaging (fMRI) Measures | 1-2 hours per session, with experiments split across multiple (e.g., 3) sessions
  7 tesla fMRI data will be acquired during visual paradigms designed to measure neural responses with and without adaptation. FMRI data will be processed and analyzed to quantify the effect of adaptation across different regions in visual cortex.
Magnetic Resonance Spectroscopy (MRS) | 1-2 hours
  7 telsa MRS data will be acquired to quantify the concentration of different brain chemicals in brain areas including visual cortex.

SECONDARY OUTCOMES:
Clinical Symptom Scores | 1-2 hours
  Measures of visual and mental symptoms, cognitive, and sensory function (e.g., Visual Snow Questionnaire), will be collected using self-report and interview methods. Scores will be compared across groups to differences in visual and mental symptoms in people with and without visual snow syndrome (VSS).

CONTACTS AND LOCATIONS:
Overall Officials: Michael-Paul Schallmo, Ph.D., Principal Investigator — University of Minnesota, Department of Psychiatry and Behavioral Sciences; Stephen A Engel, Ph.D., Study Chair — University of Minnesota, Department of Psychology; Michael S Lee, M.D., Study Chair — University of Minnesota, Department of Ophthalmology and Visual Neurosciences; Abby Metzler, M.D., Study Chair — University of Minnesota, Department of Neurology; Malgorzata Marjanska, Ph.D., Study Chair — University of Minnesota, Department of Radiology; Carrie E Robertson, M.D., Study Chair — Mayo Clinic, Rochester, Department of Neurology
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared to a public repository at the end of the study. Data that will be shared include the study protocol, informed consent form, analytic code, behavioral data, and brain imaging data.
  OpenNuero.org will be used for data and Github.com will be used to share code.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be shared within 12 months of the completion of our study or publication of a relevant manuscript, whichever comes first.
Access Criteria: Everyone will be able to access the data shared to the repositories.

REFERENCES:
- [Background] Montoya SA, Mulder CB, Allison KD, Lee MS, Engel SA, Schallmo MP. What does visual snow look like? Quantification by matching a simulation. J Vis. 2024 Jun 3;24(6):3. doi: 10.1167/jov.24.6.3. PMID 38837169
- [Background] Montoya SA, Hillstrom AJ, Allison KD, Mulder CB, Moser HR, Lee MS, Schallmo MP, Engel SA. Visual Snow Is Susceptible to the Motion Aftereffect. Invest Ophthalmol Vis Sci. 2025 Oct 1;66(13):23. doi: 10.1167/iovs.66.13.23. PMID 41085357
- [Background] Montoya SA, Mulder CB, Lee MS, Schallmo MP, Engel SA. Adapting to Visual Noise Alleviates Visual Snow. Invest Ophthalmol Vis Sci. 2023 Dec 1;64(15):23. doi: 10.1167/iovs.64.15.23. PMID 38117246
- See also: Related Info — http://schallmolab.umn.edu/